CLINICAL TRIAL: NCT02585453
Title: Influence of Lachrymal Substitute Gels on Tear Film Thickness in Patients With Moderate to Severe Dry Eye Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LT2258-PIV-0614
Record Dates: First submitted 2015-04-26; First posted 2015-10-23 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients with dry eye syndrome 1 (Experimental): 20 Patients with dry eye syndrome
  Interventions: Device: Thealoz Duo Gel
- Patients with dry eye syndrome 2 (Active Comparator): 20 Patients with dry eye syndrome
  Interventions: Device: Hylo-Gel
- Patients with dry eye syndrome 3 (Active Comparator): 20 Patients with dry eye syndrome
  Interventions: Device: Systane Gel Drops

INTERVENTIONS:
Device: Thealoz Duo Gel — Manufacturer: Laboratoires Thea, France
  Arms: Patients with dry eye syndrome 1
Device: Hylo-Gel — Manufacturer: Ursapharm, Saarbrücken, Germany
  Arms: Patients with dry eye syndrome 2
Device: Systane Gel Drops — Manufacturer: Alcon Pharma GmbH, Fort Worth, TX, USA
  Arms: Patients with dry eye syndrome 3

SUMMARY:
Dry eye syndrome is a highly prevalent ocular disease with an increasing incidence in the elderly population. Topically administered lubricants are the basis for treatment of this disease. However, exact information about the tear film thickness and the corneal residence time of topical lubricants is still sparse, therefore no ideal treatment regimen has been found.

Recently a new method for assessment of tear film thickness based on ultra high resolution optical coherence tomography (OCT) has become available. The aim of the present study is to assess tear film thickness and corneal residence time of three different formulations of topical lubricants, in particular Thealoz Duo® Eye Drops, Hylo® Gel Eye Drops and Systane® Gel Eye Drops in patients with moderate to severe dry eye disease. In addition, standard tests for dry eye syndrome, such as the ocular surface disease index (OSDI©), Schirmer I test and determination of tear break up time (BUT) will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged over 18 years
2. Signed and dated written informed consent
3. History of dry eye syndrome for at least 3 months
4. Tear Break Up Time (BUT) ≤ 10 seconds or Schirmer I test ≤ 5 mm and ≥ 2mm
5. OSDI ≥ 22
6. Normal ophthalmic findings except dry eye syndrome, ametropia < 6 Dpt.
7. No administration of topical lubricants 12-24 hours before the screening examination

Exclusion Criteria:

1. Presence of an ocular pathology judged by the investigator as incompatible with the study.
2. Any other clinical relevant ocular abnormality except DES.
3. History of allergy, known hypersensitivity to one of the components: the study medications or Fluorescein.
4. History of known clinically relevant allergy.
5. Medical or surgical history judged by the investigator to be incompatible with the study participation (hepatic or renal insufficiency; all chronic severe organic disease: metabolic, endocrine, neoplastic, haematological disease; severe psychiatric illness, etc.).
6. History of a recent acute illness with a recovery period within the 2 weeks before the inclusion visit (Day 0).
7. Pregnancy, lactation.
8. Pre-menopausal woman who is not using a reliable birth control method (oral contraceptives or coil) or is not surgically sterilised.
9. Participation in any high-speed or water-sports during the study without ocular protection (goggles or glasses).
10. Subject unable to understand the study instructions or unlikely to comply with the study schedule and treatment.
11. Participation in another clinical study in the 4 weeks before the start of the present study or at the same time as the present study.
12. Subject is a ward of court.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Tear Film thickness as measured with optical coherence tomography (OCT) | 360 minutes

SECONDARY OUTCOMES:
Tear Break Up Time | 1 month
Schirmer 1 test | 1 month
Subjective evaluation of ocular comfort | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria